CLINICAL TRIAL: NCT01778673
Title: Cortical Comminution and Intra-articular Involvement in Distal Radius Fractures Can Predict Radiological Outcome. A Prospective Multicenter Study
Status: Completed | Type: Observational
Sponsor: Sundsvall Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 09-213
Record Dates: First submitted 2013-01-24; First posted 2013-01-29 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Distal Radius Fracture; Radiological Outcome
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Distal radius fractures Sundsvall Hospital
  Interventions: Procedure: Cast immobilization
- Distal radius fractures Östersund Hospital.
  Interventions: Procedure: Cast immobilization

INTERVENTIONS:
Procedure: Cast immobilization

SUMMARY:
Background: Although fractures of the distal radius are the most common skeletal injury, the utility of the available classification systems to predict fracture stability is limited. We studied if cortical comminution and intra-articular involvement can assess instability in fractures of the distal radius.

Methods: A prospective multicenter study was conducted. Distal radius fractures in 417 skeletally mature patients (428 fractures) were studied. Fractures were divided into osteoporotic or non-osteoporotic according to age of the patients. Antero-posterior and lateral plain radiographs determined if the fractures were minimally displaced or displaced. The fracture patterns were evaluated depending on the presence and the site of cortical comminution and intra-articular involvement according to a new classification system (Buttazzoni classification). Minimally displaced fractures were treated with cast immobilization. Displaced fractures underwent closed reduction with subsequent cast immobilization. Radiographs were obtained after reduction, at 10-14 days and after 3 months. Displacement was classified as primary instability, secondary instability or late instability. Endpoints were union of the fracture or re-displacement. Results: Volarly comminuted fractures (Buttazzoni 4) displaced in 96 %, intra-articular fractures (Buttazzoni 3) in 72%, dorsally comminuted fractures (Buttazzoni 2) in 73% and non-comminuted (Buttazzoni 1) in 16 % of the cases. One third of the initially minimally displaced fractures did not maintain acceptable alignment. All initially displaced volarly comminuted fractures were unstable. In both initially displaced and minimally displaced fractures, cortical comminution and intra-articular involvement were predictive for primary, secondary and late instability.

Conclusions: Cortical comminution and intra-articular involvement seem to be valuable instruments for assessing stability at initial presentation of distal radius fractures. Level of Evidence: Level I, prospective multicenter study. Prognostic study.

DETAILED DESCRIPTION:
Between the 1st of October 2009 and the 30th of September 2011 patients with DRF at two teaching hospitals were invited to participate in a prospective study. Patients between 15 and 74 years, with closed physes of the distal radius and ulna were included. Exclusion criteria were dementia, previous fracture to the ipsilateral wrist, open fracture, other concomitant or existing damage or injury to the wrist, Galeazzi fracture, rheumatoid arthritis, alcohol or drug abuse and neurologic impairment. All patients underwent radiographic examination with frontal and lateral views centered on the wrist in neutral rotation. The radiographs were classified by the doctor on-call who had the needed information about the classification system available.

Undisplaced or minimally displaced fractures (will be called minimally displaced throughout this article) were immobilized in a Plaster-of-Paris (PoP) slab from distal to the elbow to proximal to the MCP-joints with the wrist in a neutral position. Displaced fractures were reduced under hematoma-block local anesthesia, immobilized with PoP slab and then radiologically re-examined. In cases of re-displacement at post-reduction x-ray, the fractures were registered as primary instability and further treated according to the guidelines of the treating department. Both if the fracture was minimally displaced and if reduction was successful radiographic examination was performed after 10-14 days.

If still acceptable at 10-14 days, the fractures were treated in PoP slab for totally 4-6 weeks. If the fracture at follow up had displaced, it was registered as secondary instability and further treatment was discussed. After 3 or more months radiographs were again obtained to confirm union and final position of the fracture. Fractures with an acceptable position at 10-14 days which later mal-united were registered as late instability.

If reduction to an acceptable position was not achieved initially or was lost at the 10-14 days control this was considered to be the end-point for this particular fracture in this study. Thus all fractures that entered and finished this study can either be considered to have been stable i.e. went to union in an acceptable position without operation, or were fractures that at one point or another showed that they were so unstable that an acceptable position could not be established or kept with conservative means.

Acceptable position To define acceptable and non-acceptable positions we used specific radiographic criteria. We measured volar inclination, radial tilt, ulnar variance and any eventual intra-articular step-off. It is considered that elderly people tolerate more displacement than younger people (6,10). Some authors have made an arbitrary definition, considering females above 49 years and males above 59 years as osteoporotic. Therefore; we have divided the patients into two groups, one "younger" below and one "elderly" above these ages.

For the "elderly" we accepted volar inclination up to 20°, dorsal tilt up to 10° and radial tilt of 10° or more. For the "younger" we accepted volar inclination up to 15°, dorsal tilt up to 10° and radial tilt of 15° or more. Up to 2 mm. of ulnar variance and less than 2 mm. of intra-articular step-off were acceptable in both groups.

Statistics The Fischer's exact test was used to compare each pair of class. To correct for multiple comparisons the p-values from the Fischer's exact test was corrected with Benjamini Hochberg correction. IBM SPSS 20 was used for most analysis, except for the Fischer exact with the correction where R, version 2.15 (http://www.r-project.org), was used with package fmsb. A p-value <0.05 is considered statistically significant. The false-discovery-rate for the Benjamini-Hochberg correction was set as 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients with distal radius fracture between 15 and 74 years, with closed physes of the distal radius and ulna.

Exclusion Criteria:

* Dementia, previous fracture to the ipsilateral wrist, open fracture, other concomitant or existing damage or injury to the wrist, Galeazzi fracture, rheumatoid arthritis, alcohol or drug abuse and neurologic impairment.

Ages: 15 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: community sample
Sampling Method: Probability Sample
Dates: Start 2009-10; Primary Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Fracture displacement | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of orthopedic surgery Sundsvall Hospital, Sundsvall, Sundsvall, Sweden